CLINICAL TRIAL: NCT06983925
Title: A Randomized, Open-label, Single-dose, Two-crossover Bioavailability Study of Single Oral Administration of GS1-144 Tablets Under Fasting Condition in Healthy Postmenopausal Female Subjects in China
Brief Title: A Bioavailability Study of GS1-144 Tablets in Healthy Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: GenSci074-103
Record Dates: First submitted 2025-05-06; First posted 2025-05-21 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-04

CONDITIONS: Healthy Postmenopausal Women

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- T-R (Experimental): Administration order: GS1-144 Tablet with new preparation (T), GS1-144 Tablet with present preparation (R)
  Interventions: Drug: GS1-144 Tablet with new preparation (T); Drug: GS1-144 Tablet with present preparation (R)
- R-T (Experimental): Administration order: GS1-144 Tablet with present preparation (R), GS1-144 Tablet with new preparation (T),
  Interventions: Drug: GS1-144 Tablet with new preparation (T); Drug: GS1-144 Tablet with present preparation (R)

INTERVENTIONS:
Drug: GS1-144 Tablet with new preparation (T) — GS1-144 Tablet with new preparation (T)
Drug: GS1-144 Tablet with present preparation (R) — A single oral dose of GS1-144 Tablet with present preparation

SUMMARY:
To evaluate the pharmacokinetic (PK) characteristics of GS1-144 tablets and the relative bioavailability of the two preparations in healthy postmenopausal female subjects in China.

DETAILED DESCRIPTION:
To evaluate the pharmacokinetic (PK) characteristics of GS1-144 tablets and the relative bioavailability of the two preparations in healthy postmenopausal female subjects in China.

ELIGIBILITY:
Inclusion Criteria:

* At the time of signing the Informed consent Form (ICF) : age between 40 and 65 years (inclusive of boundary values).
* Postmenopausal female subjects: Natural menopause (defined as continuous spontaneous amenorrhea for ≥ 12 months, except for lactation or surgical menopause, or continuous spontaneous amenorrhea for ≥ 6 months, serum follicle stimulating hormone (FSH) > 40 IU/L, and serum estradiol (E2) concentration less than the upper limit of the normal range in postmenopausal women; Or ≥ 6 weeks after bilateral oophorectomy (with/without hysterectomy).
* Weight ≥ 45 kg with body mass index (BMI) in the range of 18-28 kg/m2 (inclusive of boundary values).
* Be able to communicate well with researchers, understand and comply with the requirements of this study, voluntarily participate in the trial, understand and sign ICF.

Exclusion Criteria:

* (Screening/admission) Known allergic history to the study drug and any of its components or related preparations, or history of allergic diseases (including but not limited to asthma, urticaria, etc.), or allergic constitution (such as known allergic history to two or more substances).
* (Screening period/admission interrogation) Patients with any previous or current cardiovascular, gastrointestinal, endocrine, hematologic, hepatic, immunologic, metabolic, urinary, pulmonary, neurological, cutaneous, psychiatric, renal and/or other major diseases considered by the investigators as clinically significant.
* (Screening period/admission inquiry)Patients with severe infection, severe trauma or major surgical operation within 6 months before the first administration.
* (Screening period/admission inquiry) Received blood transfusion within 3 months before the first dose, or had blood donation, or had blood loss ≥400 mL, or planned to donate blood within 1 month after the end of the study.
* Abnormal detection of infectious diseases with clinical significance, such as positive human immunodeficiency virus antigen (HIV Ag) or antibody (HIV Ab), hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or treponema pallidum antibody or specific antibody.
* (Screening period/admission inquiry) Were enrolled in another clinical trial within 3 months before the first dose (except those who did not receive any intervention) or were enrolled in another clinical trial.
* (Screening period/admission inquiry) Use of any prescribed medication [including but not limited to any medication that changes liver enzyme activity (e.g., glucocorticoids, sex hormones, anticonvulsants, cyclosporine, etc.)] within 4 weeks before the first dose of medication; Or use of any non-prescription drugs (including but not limited to Chinese herbal medicine, compound preparations of Chinese herbal medicine, health supplements, etc.) and vitamin supplements within 2 weeks before administration; Those who had taken an inducer of cytochrome P450 1A2 (CYP1A2) within 3 months before taking the study drug or had taken a CYP1A2 inhibitor within the previous 2 weeks or 5 half-lives, the longer.
* Clinically significant abnormal results of physical examination, chest X-ray, abdominal ultrasound or reproductive organ ultrasound at screening; Patients with clinically significant abnormal thyroid function, parathyroid function or neck ultrasound examination results; Abnormal laboratory tests with clinical significance.
* Clinically significant abnormal vital signs, in which abnormal blood pressure was defined as systolic blood pressure ≥ 140 mmHg or < 90 mmHg, diastolic blood pressure ≥ 90 mmHg or < 60 mmHg.
* Prolonged QT interval corrected with Fridericia's formula (QTcF > 460 ms in women, Fridericia's formula: QTcF = QT/RR0.33) on 12-lead electrocardiogram at screening, or other clinically significant abnormalities.
* (Screening period/admission consultation) With a history of drug abuse at present or within 1 year.
* (Screening period/admission consultation) Smoked more than 5 cigarettes per day in the 3 months before screening, or could not stop using any tobacco products during the study period.
* (During admission) Who had a positive breath test for alcohol or had been an alcoholic for 3 months prior to screening, i.e. had consumed more than 14 units of alcohol per week (one standard unit is 17.5 mL or 14 g of pure alcohol, the alcohol content of different types of alcohol is indicated by volume, and one standard unit is approximately 35 mL of 50° liquor or 350 mL of 5° beer); Or unwilling to stop drinking alcohol or consuming any alcohol-based products during the trial.
* (During the admission period) With positive results of multiple drug tests in urine.
* (Screening period/admission inquiry) Who had consumed any food or beverage (e.g. those containing grapefruit, star fruit or their products) that might affect the metabolism of the study drug within 48 hours before admission to the phase I ward in each cycle.
* (Screening period/admission consultation) Excessive consumption (> 8 cups/day, 1 cup =250 mL) of tea, coffee or caffeinated beverages per day in the 3 months before screening; Or intake of any food or beverage (such as coffee, tea, chocolate, cola, etc.) containing or metabolized caffeine or xanthine within 24 hours before admission to phase I ward.
* Clinically significant abnormal pregnancy test results or (screening/admission inquiry) lactating women.
* Those who have difficulty in venous blood collection and/or cannot tolerate venipuncture/indwelling needle or feel dizzy with needles or blood.
* Other conditions that were considered by the investigator to be ineligible for inclusion in the trial.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2025-04-30 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (Peak Plasma Concentration (Cmax) ) of GS1-144 with present and new preparation | 0 hours -72 hours post-administration
Pharmacokinetics (Area under the blood concentration-time curve from 0 to the last quantifiable time point after administration (AUC0-t)) of GS1-144 with present and new preparation | 0 hours -72 hours post-administration
Pharmacokinetics (Area under the blood concentration-time curve from 0 to infinity (AUC0-∞)) of GS1-144 with present and new preparation | 0 hours -72 hours post-administration
Pharmacokinetics (time to peak (Tmax)) of GS1-144 with present and new preparation | 0 hours -72 hours post-administration
Pharmacokinetics (rate constant of drug elimination (λz)) of GS1-144 with present and new preparation | 0 hours -72 hours post-administration
Pharmacokinetics (elimination half-life (t1/2)) of GS1-144 with present and new preparation | 0 hours -72 hours post-administration
Pharmacokinetics (apparent clearance rate (CL/F)) of GS1-144 with present and new preparation | 0 hours -72 hours post-administration
Pharmacokinetics (apparent volume of distribution (Vz/F)) of GS1-144 with present and new preparation | 0 hours -72 hours post-administration
Pharmacokinetics (relative bioavailability (F%)) of GS1-144 with present and new preparation | 0 hours -72 hours post-administration

CONTACTS AND LOCATIONS:
Locations (1):
- Chengdu Xinhua Hospital, Chengdu, Sichuan, China